CLINICAL TRIAL: NCT01542346
Title: Subcutaneous Adaption and Cosmetic Outcome Following Caesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Klagenfurt am Wörthersee (Other)
Responsible Party: Principal Investigator, Husslein Heinrich, MD, Principal investigator, Klinikum Klagenfurt am Wörthersee
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A 16/11
Record Dates: First submitted 2012-02-25; First posted 2012-03-02 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Caesarean Delivery
Keywords: Wound closure; cosmetic outcome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (1):
- wound closure with subcutaneous adaption (Experimental)
  Interventions: Procedure: subcutaneous adaption

INTERVENTIONS:
Procedure: subcutaneous adaption

SUMMARY:
This is a double blinded randomized study investigating if subcutaneous adaption has an impact on cosmetic outcome after Caesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing cesarean section for any indication
* literate in german language

Exclusion Criteria:

* history of keloids
* previous transversal suprapubic scars
* known patient hypersensitivity to any of the suture materials used in the protocol
* a medical disorder that could affect wound healing (eg, diabetes mellitus, chronic corticosteroid use)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2012-03

PRIMARY OUTCOMES:
Objective and subjective cosmetic appearance | after 6 months

SECONDARY OUTCOMES:
Surgical site infection and wound breakdown | within 30 days after surgery
Haematoma | within 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Husslein, M.D., Principal Investigator — Klinikum Klagenfurt am Woerthersee and Medical University Vienna
Locations (1):
- Klinikum Klagenfurt am Woerthersee, Klagenfurt, Carinthia, Austria

REFERENCES:
- [Derived] Husslein H, Gutschi M, Leipold H, Herbst C, Franz M, Worda C. Suture Closure versus Non-Closure of Subcutaneous Fat and Cosmetic Outcome after Cesarean Section: A Randomized Controlled Trial. PLoS One. 2014 Dec 10;9(12):e114730. doi: 10.1371/journal.pone.0114730. eCollection 2014. PMID 25494177